CLINICAL TRIAL: NCT02291445
Title: A Randomized, Double Blind, Single Dose, Two Treatment, Two Period Crossover Pharmacokinetic Study Comparing a 182mg Colon-targeted-delivery Peppermint Oil Capsule (Tempocol-ColoPulse®) and a 182mg Enteric-coated Peppermint Oil Capsule (Tempocol®) in Healthy Volunteers
Brief Title: Comparing a 182mg Colon-targeted-delivery Peppermint Oil Capsule (Tempocol-ColoPulse®) and a 182mg Enteric-coated Peppermint Oil Capsule (Tempocol®), a Pharmacokinetic Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 50941; 2014-004195-32 (EudraCT Number)
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2015-07

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain; Colonic Diseases; Visceral Pain
Keywords: Peppermint oil; Menthol; Volatile oil; Plant oil; Visceral pain; Abdominal pain; Irritable bowel syndrome (IBS); Colonic disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Colonic Diseases; Visceral Pain | interventions — peppermint oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tempocol-ColoPulse® (Experimental): Tempocol-ColoPulse® is a colon-targeted-delivery peppermint oil capsule that will deliver peppermint oil in the (ileo-) colonic region specifically.
  Interventions: Drug: Menthae piperitae aetheroleum/peppermint oil (colon-targeted-delivery capsule)
- Tempocol® (Active Comparator): Tempocol® is an enteric-coated peppermint oil capsule that delivers peppermint oil in the upper small intestine.
  Interventions: Drug: Menthae piperitae aetheroleum/peppermint oil (enteric coated capsule)

INTERVENTIONS:
Drug: Menthae piperitae aetheroleum/peppermint oil (enteric coated capsule) — Peppermint oil capsule available as an over the counter prescription drug on the Dutch market.
  Other Names: Tempocol® (CBG-rvg number 109856)
  Arms: Tempocol®
Drug: Menthae piperitae aetheroleum/peppermint oil (colon-targeted-delivery capsule) — Peppermint oil capsule with a coating developed according to the ColoPulse® technology, ensuring a pulsatile and therefore slower release in a lower part of the intestinal tract compared to Tempocol, namely in the (ileo-)colonic region.
  Other Names: Tempocol-ColoPulse®
  Arms: Tempocol-ColoPulse®

SUMMARY:
This is a pilot study to compare the relative bioavailability between two peppermint oil formulations, namely a ileocolonic release peppermint oil and an small intestinal release peppermint oil (Tempocol®). This study is conducted as part of a future multicenter randomized controlled trial that will assess the therapeutic effect of the new peppermint oil formulation in IBS patients.

DETAILED DESCRIPTION:
Rationale: Peppermint oil has shown to be effective in the treatment of IBS symptoms in several meta-analyses. However, the level of evidence is moderate and peppermint oil remains relatively under-used in IBS. Therefore the investigators plan to conduct a multicenter randomized controlled trial to investigate the possible beneficial effects of peppermint oil in IBS. To improve efficacy and to reduce side effects, the investigators aim to study the use of a new peppermint oil formulation that will slowly release the oil in the (ileo-) colonic region specifically. In order to demonstrate differences in pharmacokinetics, the subsidizing party, ZonMW, requested an additional pilot study (described in the present protocol) in which the investigators will investigate surrogate markers for local colon bioavailability, tolerability and side effects of the new ileocolonic release PO.

Study design: a randomized, double blind, two-period, two-treatment crossover study with a wash out period of at least 14 days.

Intervention: All study volunteers will receive a single dose of 182mg of both ileocolonic release peppermint oil and small intestinal release peppermint oil, each on a different test day.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects may be confronted with certain inconveniences and minor risks. They are required to visit the MUMC+ 5 times, once for the screening and two times per test day for various non-invasive measurements (questionnaires, blood pressure and heart-rate measurement, urine and fecal sampling, pregnancy test in women in fertile ages, general physical exam) as well as for minor invasive venous blood sampling, after which a small haematoma can occur. Total time investment is +/- 30 hours, subjects will not benefit from participation.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined
* Age between 18 and 65 years
* BMI between 18 and 25 kg/m2 and a weight of at least 50 kilograms
* Women in fertile age (<55 years old) must use contraception or be postmenopausal for at least two years

Exclusion Criteria:

* History of severe or chronic cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol
* Use of medication, including vitamin and iron supplementation, except oral contraceptives, within 14 days prior to start of the study
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgment of the principle investigator)
* Dieting (for example lactose-free, gluten-free, caloric-restrictive, vegetarian or vegan, macrobiotic diet)
* Pregnancy, lactation
* High alcohol consumption (>15 alcoholic consumptions per week)
* Smoking/ Using drugs of abuse
* Self-admitted HIV-positive state
* Known allergic reaction to peppermint
* High intake of caffeine (>8 cups coffee a day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, Prof, PhD, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Maurer JM, Schellekens RC, van Rieke HM, Stellaard F, Wutzke KD, Buurman DJ, Dijkstra G, Woerdenbag HJ, Frijlink HW, Kosterink JG. ColoPulse tablets perform comparably in healthy volunteers and Crohn's patients and show no influence of food and time of food intake on bioavailability. J Control Release. 2013 Dec 28;172(3):618-24. doi: 10.1016/j.jconrel.2013.09.021. Epub 2013 Oct 2. PMID 24096020
- [Background] Schellekens RC, Stellaard F, Olsder GG, Woerdenbag HJ, Frijlink HW, Kosterink JG. Oral ileocolonic drug delivery by the colopulse-system: a bioavailability study in healthy volunteers. J Control Release. 2010 Sep 15;146(3):334-40. doi: 10.1016/j.jconrel.2010.05.028. Epub 2010 May 31. PMID 20621586
- [Background] Khanna R, MacDonald JK, Levesque BG. Peppermint oil for the treatment of irritable bowel syndrome: a systematic review and meta-analysis. J Clin Gastroenterol. 2014 Jul;48(6):505-12. doi: 10.1097/MCG.0b013e3182a88357. PMID 24100754
- [Background] Ruepert L, Quartero AO, de Wit NJ, van der Heijden GJ, Rubin G, Muris JW. Bulking agents, antispasmodics and antidepressants for the treatment of irritable bowel syndrome. Cochrane Database Syst Rev. 2011 Aug 10;2011(8):CD003460. doi: 10.1002/14651858.CD003460.pub3. PMID 21833945
- [Result] Weerts ZZRM, Keszthelyi D, Vork L, Aendekerk NCP, Frijlink HW, Brouwers JRBJ, Neef C, Jonkers DMAE, Masclee AAM. A Novel Ileocolonic Release Peppermint Oil Capsule for Treatment of Irritable Bowel Syndrome: A Phase I Study in Healthy Volunteers. Adv Ther. 2018 Nov;35(11):1965-1978. doi: 10.1007/s12325-018-0802-1. Epub 2018 Oct 4. PMID 30284674

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover design.
Groups:
- Ileocolonic Release PO First, Then Small-intestinal Release Peppermint Oil: Ileocolonic release PO is a targeted ileocolonic release peppermint oil capsule that releases peppermint oil in the (ileo-) colonic region specifically.
  Menthae piperitae aetheroleum/peppermint oil (colon-targeted-delivery capsule): Peppermint oil capsule with a coating developed according to the ColoPulse® technology, ensuring a pulsatile and therefore slower release in a lower part of the intestinal tract compared to Tempocol, namely in the (ileo-)colonic region.
- Small Intestinal Release PO First, Then Ileocolonic Release Peppermint Oil: Small Intestinal Release PO (Tempocol®) is an enteric-coated peppermint oil capsule that delivers peppermint oil in the upper small intestine.
  Menthae piperitae aetheroleum/peppermint oil (enteric coated capsule): Peppermint oil capsule available as an over the counter prescription drug on the Dutch market.
Period: Overall Study
Arm/Group | Ileocolonic Release PO First, Then Small-intestinal Release Peppermint Oil | Small Intestinal Release PO First, Then Ileocolonic Release Peppermint Oil
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ileocolonic Release PO on First Test Day: Ileocolonic release PO is a targeted ileocolonic release peppermint oil capsule that releases peppermint oil in the (ileo-) colonic region specifically.
  Menthae piperitae aetheroleum/peppermint oil (colon-targeted-delivery capsule): Peppermint oil capsule with a coating developed according to the ColoPulse® technology, ensuring a pulsatile and therefore slower release in a lower part of the intestinal tract compared to Tempocol, namely in the (ileo-)colonic region.
- Small Intestinal Release PO on First Test Day: Small Intestinal Release PO (Tempocol®) is an enteric-coated peppermint oil capsule that delivers peppermint oil in the upper small intestine.
  Menthae piperitae aetheroleum/peppermint oil (enteric coated capsule): Peppermint oil capsule available as an over the counter prescription drug on the Dutch market.
- Total: Total of all reporting groups
Arm/Group | Ileocolonic Release PO on First Test Day | Small Intestinal Release PO on First Test Day | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 21.7 [20.6 to 27.9] | 24.1 [21.2 to 55.0] | 22.2 [20.8 to 28.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 4 | 4 | 8
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 21.5 [20.6 to 22.2] | 21.7 [18.5 to 23.8] | 21.5 [20.2 to 23.0]

OUTCOME MEASURES:

1. Primary Outcome: T-max
Description: Time to reach maximum menthol-glucuronide (main constituent of peppermint oil after conversion by the liver) concentration in plasma
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Ileocolonic Release PO: Ileocolonic release PO is a targeted ileocolonic release peppermint oil capsule that releases peppermint oil in the (ileo-) colonic region specifically.
  Menthae piperitae aetheroleum/peppermint oil (colon-targeted-delivery capsule): Peppermint oil capsule with a coating developed according to the ColoPulse® technology, ensuring a pulsatile and therefore slower release in a lower part of the intestinal tract compared to Tempocol, namely in the (ileo-)colonic region.
- Small Intestinal Release PO: Small Intestinal Release PO (Tempocol®) is an enteric-coated peppermint oil capsule that delivers peppermint oil in the upper small intestine.
  Menthae piperitae aetheroleum/peppermint oil (enteric coated capsule): Peppermint oil capsule available as an over the counter prescription drug on the Dutch market.
Arm/Group | Ileocolonic Release PO | Small Intestinal Release PO
Number analyzed (Participants) | 8 | 8
minutes | 360 [360 to 405] | 180 [120 to 180]

2. Secondary Outcome: C-max
Description: Menthol-glucuronide (main constituent of peppermint oil after conversion by the liver) peak plasma concentrations
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Ileocolonic Release PO | Small Intestinal Release PO
Number analyzed (Participants) | 8 | 8
ug/L | 563.6 [268 to 849] | 702 [644 to 1020]

3. Secondary Outcome: T-lag
Description: Time until a measurable plasma concentration of menthol-glucuronide occurs after oral administration of peppermint oil (45ug/L)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Ileocolonic Release PO | Small Intestinal Release PO
Number analyzed (Participants) | 8 | 8
minutes | 225 [204 to 284] | 37 [6 to 65]

4. Secondary Outcome: AUC
Description: Area under the plasma concentration-time curve from t=0 hrs until t=24 hrs.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: ug*h/L
Arm/Group | Ileocolonic Release PO | Small Intestinal Release PO
Number analyzed (Participants) | 8 | 8
ug*h/L | 2331 [2006 to 2510] | 2623 [2471 to 2920]

5. Secondary Outcome: T1/2
Description: elimination half-life; time required for the plasma concentration of menthol-glucuronide to reach half of its original value.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ileocolonic Release PO | Small Intestinal Release PO
Number analyzed (Participants) | 8 | 8
hours | 6.1 [5.1 to 7.4] | 7.7 [7.0 to 10.8]

6. Secondary Outcome: Menthol-glucuronide Urine Exretion Time Curve
Time Frame: 24 hours
Population: No urine analysis was performed due to lack in funding. In addition, it was felt that the systemic concentration of menthol glucuronide concentration provided enough information to answer the research question.
Arm/Group | Ileocolonic Release PO First, Then Small-intestinal Release Peppermint Oil | Small Intestinal Release PO First, Then Ileocolonic Release Peppermint Oil
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: L-Menthol Concentration in Feces
Time Frame: +/- 24 hours
Reporting Status: Not Posted

8. Secondary Outcome: Difference in Total Number of Side Effects Per Time Point.
Time Frame: 24 hours
Reporting Status: Not Posted

9. Secondary Outcome: Tolerability Assessed by Heart Rate, Blood Pressure and Reported Side Effects
Description: Assessed by heart rate, blood pressure and reported side effects.
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ileocolonic Release PO | Small Intestinal Release PO
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ileocolonic Release PO (N=8) | Small Intestinal Release PO (N=8)
Acid regurgitation (Gastrointestinal disorders) | 0 | 2
Fecal urgency (Gastrointestinal disorders) | 0 | 2
Headache (General disorders) | 2 | 0
Altered Fecal Odor (Gastrointestinal disorders) | 2 | 0 — Peppermint odor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No